CLINICAL TRIAL: NCT06625814
Title: A Clinical Study to Evaluate the Effect of MK-0616 on the Pharmacokinetics of Levothyroxine in Healthy Adult Participants
Brief Title: A Study of Levothyroxine and Enlicitide Decanoate (MK-0616) in Healthy Adult Participants (MK-0616-028)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-028; MK-0616-028 (Other: MSD)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Thyroxine; MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levothyroxine (Experimental): Participants will receive a single oral dose of levothyroxine.
  Interventions: Drug: Levothyroxine
- Levothyroxine Plus Enlicitide Decanoate (Experimental): Participants will receive a single oral dose of levothyroxine and a single oral dose of enlicitide decanoate at the same time.
  Interventions: Drug: Levothyroxine; Drug: Enlicitide Decanoate

INTERVENTIONS:
Drug: Levothyroxine — single oral dose
  Other Names: Synthroid
Drug: Enlicitide Decanoate — single oral dose
  Other Names: MK-0616
  Arms: Levothyroxine Plus Enlicitide Decanoate

SUMMARY:
Levothyroxine (T4) is a man-made thyroid hormone used to treat certain thyroid conditions. After taking levothyroxine, a person's body changes it to triiodothyronine (T3). The amount of levothyroxine in a person's blood must be carefully controlled to maintain proper function. Enlicitide decanoate was designed to lower the amount of cholesterol in a person's blood.

Researchers want to learn about levothyroxine when taken at the same time with enlicitide decanoate. They want to:

* Measure a person's blood to find out if the amount of levothyroxine in the blood is the same when levothyroxine is taken alone or with enlicitide decanoate
* Learn about the safety of levothyroxine when taken alone or with enlicitide decanoate and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Medically healthy with no clinically significant medical history
* Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* History of cardiovascular disease or diabetes mellitus
* History of cancer

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve from Time 0 to 48 hours (AUC0-48hrs) of Levothyroxine (total T4) | At designated timepoints (up to approximately 48 hours postdose)
  Blood samples will be collected to determine the AUC0-48hr of Levothyroxine (T4).
Maximum Plasma Concentration (Cmax) of Levothyroxine (total T4) | At designated timepoints (up to approximately 48 hours postdose)
  Blood samples will be collected to determine the Cmax of Levothyroxine (T4).
Time to Maximum Plasma Concentration (Tmax) of Levothyroxine (total T4) | At designated timepoints (up to approximately 48 hours postdose)
  Blood samples will be collected to determine the Tmax of Levothyroxine (T4).
Area under the Concentration-Time Curve from Time 0 to 48 hours (AUC0-48hrs) of Triiodothyronine (total T3) | At designated timepoints (up to approximately 48 hours postdose)
  Blood samples will be collected to determine the AUC0-48hr of triiodothyronine (T3).
Maximum Plasma Concentration (Cmax) of Triiodothyronine (total T3) | At designated timepoints (up to approximately 48 hours postdose)
  Blood samples will be collected to determine the Cmax of triiodothyronine (T3).
Time to Maximum Plasma Concentration (Tmax) of Triiodothyronine (total T3) | At designated timepoints (up to approximately 48 hours postdose)
  Blood samples will be collected to determine the Tmax of triiodothyronine (T3).

SECONDARY OUTCOMES:
Number of Participants Who Experience a Treatment-Emergent Adverse Event (TEAE) | Up to approximately 7 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE will be considered treatment-emergent if the onset date and time is at the time of or after the first study drug administration. The number of participants who experience a TEAE will be reported.
Number of Participants Who Discontinue Study Due to a TEAE | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE will be considered treatment-emergent if the onset date and time is at the time of or after the first study drug administration. The number of participants who discontinue study due to a TEAE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com